CLINICAL TRIAL: NCT06409793
Title: Motivating Adolescent Fitness
Acronym: MOTAFIT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: MOSS ROCK PARK FOUNDATION (Unknown)
Responsible Party: Principal Investigator, Ai McManus, Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: UBC MOTAFIT
Record Dates: First submitted 2024-03-04; First posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Exercise Training
MeSH Terms: interventions — Telemedicine

STUDY DESIGN:
Intervention Model Description: The proposed intervention will provide one group of adolescents with a combined accelerometer and heart rate monitor, alongside exercise counselling. The accelerometer will be used to support the youngsters achieve a personalised daily PA goal. The heart rate monitor will then be used to support adherence to an individualised and co-created home-based exercise programme.
  A second group will receive exercise counselling only.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- mHealth (Experimental): Participants will undertake a 3-month structured exercise and PA intervention, supported by an exercise specialist. Participants will have 5 exercise consultations. Participants will receive a personalised progressive exercise programme. The aim will be to increase exercise intensity and duration during the first 3-months; aiming to meet the aerobic training guidelines of 3-4 sessions of at least 40 minutes at 85-90% heart rate maximum or of vigorous intensity. During follow-up, the aim will be to at least maintain this level of exercise.
  Participants will receive 1) a wrist worn fitness watch (Polar Ignite), featuring a 3d accelerometer and optical heart rate monitor, and 2) a smartphone app for participants (Polar Flow - Sync & Analyse). These will be synced, allowing data to be transferred to the exercise specialist, who will created monitor pre-set exercise sessions.
  Interventions: Behavioral: mHealth
- Exercise Counselling (Active Comparator): Participants will undertake the same 3-month structured exercise and PA intervention, supported by an exercise specialist, but without the use of mHealth technology to support the prescription and adherence to the exercise.
  Participants will be monitored using a wrist worn fitness watch, but will not receive feedback or have pre-set exercise sessions through the mHealth technology
  Interventions: Behavioral: mHealth
- Active control (No Intervention): Participants will receive no exercise or PA intervention. Participants will continue with regular PA behaviours as an active control comparator. Participants in the control group will be monitored at the start and the end of the 3 months intervention period (2 weeks) to determine habitual PA and exercise levels

INTERVENTIONS:
Behavioral: mHealth — A 3-month structured exercise and PA intervention, supported by an exercise specialist, with a 3-month follow-up
  Other Names: Exercise Counselling
  Arms: Exercise Counselling; mHealth

SUMMARY:
The researchers are investigating whether adding mobile technology to a home-based exercise counselling program makes it easier for youth to begin and maintain regular exercise. Participants who joins the study will receive exercise counselling from an exercise specialist, but half of all participants will receive mobile technology - a fitness watch - that links to a mobile phone App. The mobile App allows the exercise specialist to provide personalized feedback throughout the program via the fitness watch. The investigators are interested to know whether the fitness watch and mobile App will make it easier for youth to achieve their exercise goals. Both groups will be compared to an active control group, who will receive no exercise program.

DETAILED DESCRIPTION:
Purpose:

The investigators aim to undertake an experimental trial using exercise training in adolescents, evaluating a theoretical model where mHealth technology, allowing biometric informed feedback and coaching, is incorporated into a structured home-based exercise and physical activity (PA) intervention. The overall objective is to have an evidence-based exercise and PA intervention ready to evaluate in a future randomised controlled trial (RCT).

Hypothesis:

It is hypothesized that this approach will increase both habitual PA and adherence to structured exercise of the appropriate intensity to promote improvements in cardiorespiratory fitness and vascular function.

Justification:

Current physical activity guidelines suggest adolescents should accumulate at least 60 minutes of moderate to vigorous physical activity (MVPA) per day. Yet globally, more than 80% of adolescents fail to achieve the recommended level of daily MVPA, and less than 25% of Canadian adolescents are sufficiently physically active. Adolescence is a time when sedentary habits predominantly manifest. Sedentary time increases by approximately 100 minutes/day between the ages 12 and 16 years, and there is a disproportionate number of inactive adolescent girls (82%) compared to boys (71%). Clearly current strategies to encourage appropriate levels of physical activity in adolescence are inadequate.

It is important to note that the current MVPA guidelines lack the intensity associated with the enhancement of cardiorespiratory fitness in youth (~85-90% of heart rate maximum).Further, the extant data show that habitual physical activity is not related, or at best weakly related to direct laboratory measures of cardiorespiratory fitness in youth.

If we aspire to improve cardiorespiratory or vascular health in our younger population, we need to find ways to engage adolescents in sufficient exercise i.e., 40-60 minutes, 3 to 4 times per week at ~85-90% of heart rate maximum.

Objectives:

Primary Objective

1) Determine the number of sedentary adolescents that are eligible to participate, the proportion of these who would be willing to take part in this trial, and their characteristics, and the number of participants retained at 6-months.

Secondary Objectives

1. Adherence to the exercise training.
2. Estimate precision of potential outcome measures required for sample size estimations for the definitive RCT.
3. Intervention acceptability

Research Design:

The study is a randomised controlled intervention, whereby participants will complete pre-randomisation baseline testing (T1) before a 3-month supported PA and exercise intervention is completed. Immediately post-intervention (T2) and 6-months after the intervention is completed

Statistical Analysis:

The proportion of eligible patients who consent to participate in the pilot will be presented, along with the proportions in each intervention group completing each follow up assessment and the reasons for withdrawal. Descriptive characteristics and outcome data will be summarized overall and by intervention group, as mean (standard deviation) for normally distributed continuous variables, median (interquartile range) for non-normally distributed continuous variables, and number (percentage) for categorical variables.

Interview data will be analysed using thematic analysis, which will allow the research team to discuss emerging themes and help the research team to explore the barriers and facilitators to the intervention and refine the theoretical model, assessing which elements of the intervention. are most effective for participants. As this is a pilot study there will be no formal comparisons between groups in the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Aged 13-16 years
* Be comfortable communicating in English

Exclusion Criteria:

* Aged <13 or >16
* Inability to increase level of activity or exercise
* Not owning a smartphone/ or having no data plan or access to Wi-Fi
* Currently meeting the recommended exercise guidelines
* Have congenital cardiac abnormalities (e.g., tetralogy of Fallot)
* Have a known respiratory disease (e.g., asthma)
* Have a known metabolic disease (e.g., Type 1 diabetes)
* Are pregnant

Ages: 13 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Eligibility to participate in the intervention | Baseline, and follow up at weeks 4,8,12
  1. The number of adolescents approached and reasons for not joining the study
  2. Number of participants approached to participate, percentage attending/ dropout throughout the intervention
Enrolment in the intervention | Baseline, week 12
  Percentage of adolescents attending at 3-month post and 6-month follow up and reasons for drop-out.

SECONDARY OUTCOMES:
Adherence | 12 weeks
  Adherence to the exercise training. Assessed as the number of prescribed sessions completed (as a percentage), and as the percentage of each exercise session spent in desired heart rate zones (80-95% heart rate max).
Precision of potential outcome measures of cardiorespiratory fitness | Baseline, week 12, week 24
  Estimate precision of potential outcome measures required for sample size estimations for the definitive RCT. Maximal oxygen uptake will be assessed on an bike ergometer ramp incremental test to exhaustion. This will be compared from pre compared to post intervention
Precision of potential outcome measures of peripheral vascular function | Baseline, week 12, week 24
  Estimate precision of potential outcome measures required for sample size estimations for the definitive RCT. This is assessed using ultrasound to assess peripheral endothelial function of the brachial artery at baseline compared to post intervention and follow up assessment.
Precision of potential outcome measures of cerebrovascular function | Baseline, week 12, week 24
  Cerebrovascular function will be assessed using ultrasound of the internal carotid artery and vertebral artery for measures of blood flow and shear rate. This will be compared from baseline to post intervention.
Acceptability of the exercise training program | baseline, week 6 and week 12
  This will be assessed using validated PACES 5-point likert scales for enjoyment of exercise sessions, self efficacy, positive and negative affect and perceived behavioural control. These will be assessed on a 5 point scale from 1-5 of participants subjective feelings throughout the intervention, and compared to participants between different arms of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Alison McManus, PhD, Principal Investigator — University of British Columbia- Okanagan
Locations (1):
- University of British Columbia, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
The data collected will be kept by Dr McManus and Dr Koep and written up for publication

REFERENCES:
- [Derived] Koep JL, Sansum KM, Low J, Smith KJ, Cocks M, McManus AM. Feasibility of a mobile health intervention to motivate adolescent fitness and high-intensity exercise adherence (Motivating Adolescent Fitness (MOTAFIT)): protocol for a randomised controlled trial. BMJ Open. 2026 Feb 10;16(2):e112546. doi: 10.1136/bmjopen-2025-112546. PMID 41667175